CLINICAL TRIAL: NCT02479724
Title: A-line/CareTaker Comparison Study in ICU Patients
Status: Completed | Type: Observational
Sponsor: Empirical Technologies Corporation (Industry)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Other Study IDs: ETC_CareTaker_01
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Blood Pressure
Keywords: continuous, non-invasive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: continuous non-invasive blood pressure monitor — continuous blood pressure monitoring using device in parallel with Gold Standard (A-line)

SUMMARY:
Comparison of Blood Pressures obtained with the Pulse Decomposition Algorithm and Intra-Arterial Catheters in ICU Patients

DETAILED DESCRIPTION:
The object of the work presented here was to validate a new approach to tracking blood pressure that is based on the pulse analysis of the peripheral arterial pressure pulse. The approach, referred to as the Pulse Decomposition Analysis (PDA) model, goes beyond traditional pulse analysis by invoking a physical model that comprehensively links the components of the peripheral pressure pulse envelope with two reflection sites in the central arteries.

In these experiments, approved by the University of Virginia Institutional Review Board, the arterial blood pressures of patients (23 m/11 f, mean age: 44.05 y, SD: 13.9 y, mean height: 173.3 cm, SD: 9.4 cm, mean weight: 95.3 kg, SD: 27.4 kg) hospitalized in University of Virginia Medical Intensive Care Units (MICUs) were monitored using radial intra-arterial catheters, while the CareTaker system collected pulse line shapes at the lower phalange of the thumb of the ipsilateral hand.

Systolic and diastolic blood pressures continuously collected from the arterial catheter and CT were compared. Pearson correlation coefficients were calculated between arterial catheter and CT blood pressure measurements and a Bland-Altman analysis was created. Results were within the limits established for the validation of automatic arterial pressure monitoring (AAMI/ANSI/ISO 81060-1:2013).

ELIGIBILITY:
Inclusion Criteria:

* male or female age 18 to 45
* presence of a radial arterial catheter
* informed consent by subject or surrogate
* available digital pulse

Exclusion Criteria:

* failure to meet all of the inclusion criteria

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: (23 m/11 f, mean age: 44.05 y, SD: 13.9 y, mean height: 173.3 cm, SD: 9.4 cm, mean weight: 95.3 kg, SD: 27.4 kg) hospitalized in University of Virginia Medical Intensive Care Units (MICUs)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Performance comparison according to AAMI/ANSI/ISO 81060-1:2013 | 40 minutes
  Correlation and standard deviation between both blood pressure measurement systems were assessed according to 81060 standards.

CONTACTS AND LOCATIONS:
Overall Officials: Martin C. Baruch, PhD, Principal Investigator — Empirical Technologies Corporation